CLINICAL TRIAL: NCT06192004
Title: An Observational, Prospective, Multicenter Study of Non-Small Cell Lung Cancer Patients in the US Receiving Standard-of-Care and Initiating an Approved Therapy With Risk of Pneumonitis/ILD
Brief Title: Study of Non-Small Cell Lung Cancer Patients in the US Receiving Standard-of-Care and Initiating an Approved Therapy With Risk of Pneumonitis/ILD
Acronym: LOOP
Status: Terminated | Type: Observational
Why Stopped: Observed event rate was below the rate required to meet study objectives.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7680C00001
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Standard-of-Care; pneumonitis; Interstitial lung disease (ILD)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pneumonia; Lung Diseases, Interstitial | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: NSCLC patients initiating an approved treatment with risk of pneumonitis/ILD.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — Not applicable since Observational Study
  Other Names: Observational Study

SUMMARY:
This is an observational, prospective, multicenter study conducted in the US to gather evidence in the context of lung cancer to complement the development of a digital solution.

Patients initiating treatment for non-small cell lung cancer (NSCLC) will be prospectively followed to characterize risk factors, signs, and symptoms leading to onset, diagnosis, and treatment of pneumonitis/ILD should it occur.

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter study conducted in the US to gather evidence in the context of lung cancer to complement the development of a digital solution.

Data will be collected prospectively from study sites using eCRFs and remotely from patients using a digital health tool.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or older, at the time of signing the ICF (Informed consent).
2. Have histologically or cytologically documented unresectable Stage III or Stage IV NSCLC.
3. Are initiating treatment with an FDA (Food and Drug Administration)-approved immune checkpoint inhibitor (alone or in combination with other agents), antibody drug conjugate, or small molecule EGFR inhibitor.
4. Minimum life expectancy of 12 weeks at the time of signing the ICF.
5. Able and willing to provide written signed informed consent.
6. Able and willing to use the digital health tool throughout the duration of the study.

Exclusion Criteria:

1. Concurrent participation in a research study or a clinical trial.
2. Unable to receive SoC for the treatment and management of NSCLC including clinical or imaging assessments for up to 6 months.
3. Judgment by the Investigator that the patient is unsuitable to participate in the study and/or the patient is unlikely to comply with study procedures and requirements.
4. Confirmed or suspected diagnosis of pneumonitis/ILD at the time of signing ICF. This does not apply to historical pneumonitis/ILD events that have resolved prior to signing ICF.
5. More than 2 weeks have passed from the administration of the first dose of qualifying FDA-approved treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients initiating an approved treatment with risk of pneumonitis/ILD; receiving SoC and initiating treatment with an FDA-approved immune checkpoint inhibitor (alone or in combination with other agents), antibody drug conjugate, or small molecule EGFR inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity, Specificity, positive predictive value (PPV), negative predictive value (NPV) and odds ratio (OR) of the algorithm | Approximately 6 months
  To complement the development of the algorithm to identify a patient at risk of pneumonitis/ILD.

SECONDARY OUTCOMES:
Sensitivity, specificity, PPV, NPV and OR of the algorithm | Approximately 6 months
  To assess algorithm performance in identifying Pneumonitis/ILD and other lung/respiratory/thoracic-related events including but not limited to: tumor progression, pneumonia, COVID-19.
Incidence of pneumonitis/ILD per grade | Approximately 6 months
  To characterize the onset and evolution over time of pneumonitis/ILD in patient receiving SoC for NSCLC.
Time from anti-tumor treatment initiation to suspicion of pneumonitis/ILD | Approximately 6 months
  To characterize the onset and evolution over time of pneumonitis/ILD in patient receiving SoC for NSCLC.
Time from anti-tumor treatment initiation to pneumonitis-related anti-tumor treatment dose delay, dose reduction, and/or discontinuation | Approximately 6 months
  To characterize the onset and evolution over time of pneumonitis/ILD in patient receiving SoC for NSCLC.
Time from pneumonitis-related treatment or diagnosis to anti-tumor treatment dose delay, dose reduction, and/or discontinuation | Approximately 6 months
  To characterize the onset and evolution over time of pneumonitis/ILD in patient receiving SoC for NSCLC.
Time from pneumonitis-related anti-tumor treatment discontinuation to rechallenge | Approximately 6 months
  To characterize the onset and evolution over time of pneumonitis/ILD in patient receiving SoC for NSCLC.
Resources used for the monitoring, diagnosis, or management of pneumonitis/ILD | Approximately 6 months
  The use of corticosteroids, test(s) requirements for diagnosis, hospitalization will be evaluated to characterize the onset and evolution over time of pneumonitis/ILD in patient.
Change from baseline in St George's Respiratory Questionnaire (SGRQ-I) health status score | Approximately 6 months
  St George's Respiratory Questionnaire for Idiopathic Pulmonary Fibrosis
Change from baseline in 5 Level EuroQoL 5 Dimension Questionnaire (EQ-5D-5L) health status score | Approximately 6 months
  5 Level EuroQoL 5 Dimension Questionnaire
Change from baseline in symptom severity score | Approximately 6 months
  Daily symptom severity rating
Compliance rate of patient-reported symptoms | Approximately 6 months
  Daily symptom severity rating
Compliance rate of patient collected pulse oximetry assessment | Approximately 6 months
  Daily pulse oximetry reading
Incidence of pneumonitis/ILD and other lung/respiratory/thoracic-related events | Approximately 6 months
  The incidence of pneumonitis/ILD and other lung/respiratory/thoracic-related events including but not limited to tumor progression, pneumonia, COVID-19, and associations and correlations with patient-generated data on eCOA will be assessed.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Miami Lakes, Florida
  - Research Site, Skokie, Illinois
  - Research Site, Ames, Iowa
  - Research Site, Covington, Louisiana
  - Research Site, Troy, Michigan
  - Research Site, Florham Park, New Jersey
  - Research Site, Mickleton, New Jersey
  - Research Site, Shirley, New York
  - Research Site, Westbury, New York
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, York, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Longview, Texas
  - Research Site, Odessa, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/